CLINICAL TRIAL: NCT02844374
Title: Epileptogenic Zone's Cartography by Quantification of EEG's Signal and Intracerebral Stimulation.
Acronym: EPISTIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 38RC14.079
Record Dates: First submitted 2016-07-18; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Epilepsy
Keywords: Epilepsy; Surgery candidate; EEG's Signal
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Partial Epilepsy Drug Resistant (Other): Patients with partial Epilepsy Drug Resistant , justifying a SEEG exploration.
  Interventions: Other: Functional stereotaxic exploration

INTERVENTIONS:
Other: Functional stereotaxic exploration — Visual analysis : in order to define the level of cortical resections. Epileptogenic maps : calculated for each crisis and for all crisis in general. Connectivity maps : calculated for each site stimulated at low-frequency. Post-operative evaluation : in order to assess the extent of resection.
  Other Names: sEEG

SUMMARY:
Epilepsy is a devastating chronic disease due to multiple causes that affect close to 50% of the world's population.

Although effective, epilepsy surgery fails in many cases, the percentage of patients free from crisis on a long term (≥ 5 years) varies from 27% to 66% according to the kind of epilepsy.

It is in this context that EPISTIM is interesting, and its aims isb a better electrophysiology delimiting of cortical networks that imply the genesis of seizures with the aim to improove surgery results.

This study will rely on the intracerebral records and on corticales electrical stimulation as they are currently routinely used by epileptic patients candidates for surgery.

ELIGIBILITY:
Inclusion Criteria :

* Patient from 5 to 65 years (L1121-7 L1122 2 CSP), including legally protected or unable to give his consent (L1121-8 CSP).
* Written approval of inclusion in the study from the patient or his legal representative.
* Patients with partial Epilepsy Drug Resistant , justifying a SEEG exploration.

Exclusion Criteria :

* Patient under 5 years.
* Patient over 65 years.
* Pregnant or breastfeeeding women (L1121-5 CSP).
* Patient deprived of liberty as a result of a judicial or administrative decision (L1121-6 CSP).
* Patients over 18 years unable to give their free consent and not subject to a legal protection order.

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Visual analysis | up to one hour
  Visual analysis : in order to define the level of cortical resections.
Epileptogenic maps | up to 10 min
  Epileptogenic maps : calculated for each crisis and for all crisis in general.
Connectivity maps | up to 10 min
  Connectivity maps : calculated for each site stimulated at low-frequency.
MRI | up to one hour
  Post-operative evaluation : in order to assess the extent of resection. MRI : 3D-T1

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Kahane, Professor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Alarcon G, Binnie CD, Elwes RD, Polkey CE. Power spectrum and intracranial EEG patterns at seizure onset in partial epilepsy. Electroencephalogr Clin Neurophysiol. 1995 May;94(5):326-37. doi: 10.1016/0013-4694(94)00286-t. PMID 7774519
- [Background] Allen PJ, Fish DR, Smith SJ. Very high-frequency rhythmic activity during SEEG suppression in frontal lobe epilepsy. Electroencephalogr Clin Neurophysiol. 1992 Feb;82(2):155-9. doi: 10.1016/0013-4694(92)90160-j. PMID 1370786
- [Background] Bartolomei F, Chauvel P, Wendling F. Epileptogenicity of brain structures in human temporal lobe epilepsy: a quantified study from intracerebral EEG. Brain. 2008 Jul;131(Pt 7):1818-30. doi: 10.1093/brain/awn111. Epub 2008 Jun 13. PMID 18556663
- [Background] Blauwblomme T, Kahane P, Minotti L, Grouiller F, Krainik A, Vercueil L, Chabardes S, Hoffmann D, David O. Multimodal imaging reveals the role of gamma activity in eating-reflex seizures. J Neurol Neurosurg Psychiatry. 2011 Oct;82(10):1171-3. doi: 10.1136/jnnp.2010.212696. Epub 2010 Nov 19. PMID 21097547
- [Background] Bulacio JC, Jehi L, Wong C, Gonzalez-Martinez J, Kotagal P, Nair D, Najm I, Bingaman W. Long-term seizure outcome after resective surgery in patients evaluated with intracranial electrodes. Epilepsia. 2012 Oct;53(10):1722-30. doi: 10.1111/j.1528-1167.2012.03633.x. Epub 2012 Aug 20. PMID 22905787
- [Background] Cossu M, Cardinale F, Castana L, Citterio A, Francione S, Tassi L, Benabid AL, Lo Russo G. Stereoelectroencephalography in the presurgical evaluation of focal epilepsy: a retrospective analysis of 215 procedures. Neurosurgery. 2005 Oct;57(4):706-18; discussion 706-18. PMID 16239883
- [Background] Catenoix H, Magnin M, Guenot M, Isnard J, Mauguiere F, Ryvlin P. Hippocampal-orbitofrontal connectivity in human: an electrical stimulation study. Clin Neurophysiol. 2005 Aug;116(8):1779-84. doi: 10.1016/j.clinph.2005.03.016. PMID 16002335
- [Background] Catenoix H, Magnin M, Mauguiere F, Ryvlin P. Evoked potential study of hippocampal efferent projections in the human brain. Clin Neurophysiol. 2011 Dec;122(12):2488-97. doi: 10.1016/j.clinph.2011.05.007. Epub 2011 Jun 12. PMID 21669549
- [Background] David O, Bastin J, Chabardes S, Minotti L, Kahane P. Studying network mechanisms using intracranial stimulation in epileptic patients. Front Syst Neurosci. 2010 Oct 20;4:148. doi: 10.3389/fnsys.2010.00148. eCollection 2010. PMID 21060722
- [Background] David O, Blauwblomme T, Job AS, Chabardes S, Hoffmann D, Minotti L, Kahane P. Imaging the seizure onset zone with stereo-electroencephalography. Brain. 2011 Oct;134(Pt 10):2898-911. doi: 10.1093/brain/awr238. PMID 21975587
- [Background] Engel J Jr, Van Ness Paul C, Rasmussen TB, Ojemann LM. Outcome with respect to epileptic seizures. In: Engel J Jr, editor. Surgical treatment of the epilepsies, 2d ed. Philadelphia: Lippincott-Raven; 1996: 609-621.
- [Background] Fisher RS, Webber WR, Lesser RP, Arroyo S, Uematsu S. High-frequency EEG activity at the start of seizures. J Clin Neurophysiol. 1992 Jul;9(3):441-8. doi: 10.1097/00004691-199207010-00012. PMID 1517412
- [Background] Gordon B, Lesser RP, Rance NE, Hart J Jr, Webber R, Uematsu S, Fisher RS. Parameters for direct cortical electrical stimulation in the human: histopathologic confirmation. Electroencephalogr Clin Neurophysiol. 1990 May;75(5):371-7. doi: 10.1016/0013-4694(90)90082-u. PMID 1692272
- [Background] Jallon P. [Epidemiology of drug-resistant epilepsies]. Rev Neurol (Paris). 2004 Jun;160 Spec No 1:5S22-30. French. PMID 15331944
- [Background] Jirsch JD, Urrestarazu E, LeVan P, Olivier A, Dubeau F, Gotman J. High-frequency oscillations during human focal seizures. Brain. 2006 Jun;129(Pt 6):1593-608. doi: 10.1093/brain/awl085. Epub 2006 Apr 21. PMID 16632553
- [Background] Kahane P, Bartolomei F. Traitement neurochirurgical de l'épilepsie. EMC (Elsevier Masson SAS, Paris), Neurologie, 17-045-A-53, 2011.
- [Background] Kahane P, Tassi L, Francione S, Hoffmann D, Lo Russo G, Munari C. [Electroclinical manifestations elicited by intracerebral electric stimulation "shocks" in temporal lobe epilepsy]. Neurophysiol Clin. 1993 Jul;23(4):305-26. doi: 10.1016/s0987-7053(05)80123-6. French. PMID 8332107
- [Background] Kahane P, Minotti L, Hoffmann D, Lachaux JP, Ryvlin P. Invasive EEG in the definition of the seizure onset zone: depth electrodes. In : Rosenow F, Lüders HO, eds. Handbook of Clinical Neurophysiology, Vol.3. Presurgical assessment of the epilepsies with clinical neurophysiology and functional imaging. Amsterdam : Elsevier BV, 2004 : 109-133.
- [Background] Kahane P, Ryvlin P, Vercueil L, Hirsch E, Arzimanoglou A. [In this era of value for money what is the place of epilepsy surgery in hospital practice]. Rev Neurol (Paris). 2007 Dec;163(12):1151-6. doi: 10.1016/S0035-3787(07)78399-6. No abstract available. French. PMID 18355462
- [Background] Koubeissi MZ, Lesser RP, Sinai A, Gaillard WD, Franaszczuk PJ, Crone NE. Connectivity between perisylvian and bilateral basal temporal cortices. Cereb Cortex. 2012 Apr;22(4):918-25. doi: 10.1093/cercor/bhr163. Epub 2011 Jun 29. PMID 21715651
- [Background] Kwan P, Brodie MJ. Early identification of refractory epilepsy. N Engl J Med. 2000 Feb 3;342(5):314-9. doi: 10.1056/NEJM200002033420503. PMID 10660394
- [Background] Lacruz ME, Garcia Seoane JJ, Valentin A, Selway R, Alarcon G. Frontal and temporal functional connections of the living human brain. Eur J Neurosci. 2007 Sep;26(5):1357-70. doi: 10.1111/j.1460-9568.2007.05730.x. PMID 17767512
- [Background] Lee SA, Spencer DD, Spencer SS. Intracranial EEG seizure-onset patterns in neocortical epilepsy. Epilepsia. 2000 Mar;41(3):297-307. doi: 10.1111/j.1528-1157.2000.tb00159.x. PMID 10714401
- [Background] Matsumoto R, Nair DR, LaPresto E, Najm I, Bingaman W, Shibasaki H, Luders HO. Functional connectivity in the human language system: a cortico-cortical evoked potential study. Brain. 2004 Oct;127(Pt 10):2316-30. doi: 10.1093/brain/awh246. Epub 2004 Jul 21. PMID 15269116
- [Background] Matsumoto R, Nair DR, LaPresto E, Bingaman W, Shibasaki H, Luders HO. Functional connectivity in human cortical motor system: a cortico-cortical evoked potential study. Brain. 2007 Jan;130(Pt 1):181-97. doi: 10.1093/brain/awl257. Epub 2006 Oct 17. PMID 17046857
- [Background] Matsumoto R, Nair DR, Ikeda A, Fumuro T, Lapresto E, Mikuni N, Bingaman W, Miyamoto S, Fukuyama H, Takahashi R, Najm I, Shibasaki H, Luders HO. Parieto-frontal network in humans studied by cortico-cortical evoked potential. Hum Brain Mapp. 2012 Dec;33(12):2856-72. doi: 10.1002/hbm.21407. Epub 2011 Sep 19. PMID 21928311
- [Background] Morris H, Najm I, Kahane P. Epilepsy surgery : patient selection. In: Lüders HO, ed. Textbook of epilepsy surgery. London : Informa Healthcare, 2008: 230-237.
- [Background] Munari C, Bancaud J. The role of stereo-electro-encephalography (SEEG) in the evaluation of partial epileptic patients. In: Porter RJ, Morselli PL, eds. The epilepsies. London : Butterworths, 1987 : 267-306.
- [Background] Nariai H, Nagasawa T, Juhasz C, Sood S, Chugani HT, Asano E. Statistical mapping of ictal high-frequency oscillations in epileptic spasms. Epilepsia. 2011 Jan;52(1):63-74. doi: 10.1111/j.1528-1167.2010.02786.x. Epub 2010 Nov 18. PMID 21087245
- [Background] Nathan SS, Sinha SR, Gordon B, Lesser RP, Thakor NV. Determination of current density distributions generated by electrical stimulation of the human cerebral cortex. Electroencephalogr Clin Neurophysiol. 1993 Mar;86(3):183-92. doi: 10.1016/0013-4694(93)90006-h. PMID 7680994
- [Background] Ochi A, Otsubo H, Donner EJ, Elliott I, Iwata R, Funaki T, Akizuki Y, Akiyama T, Imai K, Rutka JT, Snead OC 3rd. Dynamic changes of ictal high-frequency oscillations in neocortical epilepsy: using multiple band frequency analysis. Epilepsia. 2007 Feb;48(2):286-96. doi: 10.1111/j.1528-1167.2007.00923.x. PMID 17295622
- [Background] Penfield W, Jasper H, eds. Epilepsy and the functional anatomy of the human brain. Boston: Little, Brown and Company, 1954.
- [Background] Picot MC, Baldy-Moulinier M, Daures JP, Dujols P, Crespel A. The prevalence of epilepsy and pharmacoresistant epilepsy in adults: a population-based study in a Western European country. Epilepsia. 2008 Jul;49(7):1230-8. doi: 10.1111/j.1528-1167.2008.01579.x. PMID 18363709
- [Background] Rosenberg DS, Mauguiere F, Catenoix H, Faillenot I, Magnin M. Reciprocal thalamocortical connectivity of the medial pulvinar: a depth stimulation and evoked potential study in human brain. Cereb Cortex. 2009 Jun;19(6):1462-73. doi: 10.1093/cercor/bhn185. Epub 2008 Oct 20. PMID 18936272
- [Background] Schmidt D, Baumgartner C, Loscher W. The chance of cure following surgery for drug-resistant temporal lobe epilepsy. What do we know and do we need to revise our expectations? Epilepsy Res. 2004 Jul-Aug;60(2-3):187-201. doi: 10.1016/j.eplepsyres.2004.07.004. PMID 15380563
- [Background] Tellez-Zenteno JF, Dhar R, Wiebe S. Long-term seizure outcomes following epilepsy surgery: a systematic review and meta-analysis. Brain. 2005 May;128(Pt 5):1188-98. doi: 10.1093/brain/awh449. Epub 2005 Mar 9. PMID 15758038
- [Background] Valentin A, Anderson M, Alarcon G, Seoane JJ, Selway R, Binnie CD, Polkey CE. Responses to single pulse electrical stimulation identify epileptogenesis in the human brain in vivo. Brain. 2002 Aug;125(Pt 8):1709-18. doi: 10.1093/brain/awf187. PMID 12135963
- [Background] Wendling F, Bartolomei F, Bellanger JJ, Bourien J, Chauvel P. Epileptic fast intracerebral EEG activity: evidence for spatial decorrelation at seizure onset. Brain. 2003 Jun;126(Pt 6):1449-59. doi: 10.1093/brain/awg144. PMID 12764064
- [Background] Wilson CL, Isokawa M, Babb TL, Crandall PH. Functional connections in the human temporal lobe. I. Analysis of limbic system pathways using neuronal responses evoked by electrical stimulation. Exp Brain Res. 1990;82(2):279-92. doi: 10.1007/BF00231248. PMID 2286232
- [Background] Worrell GA, Parish L, Cranstoun SD, Jonas R, Baltuch G, Litt B. High-frequency oscillations and seizure generation in neocortical epilepsy. Brain. 2004 Jul;127(Pt 7):1496-506. doi: 10.1093/brain/awh149. Epub 2004 May 20. PMID 15155522